CLINICAL TRIAL: NCT01819493
Title: Parents and Children Together Preventing Diabetes
Brief Title: Parents and Children Together Preventing Diabetes (PACT PD)
Acronym: PACT PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00021267; R34DK094108-01A1 (NIH)
Record Dates: First submitted 2013-03-22; First posted 2013-03-27 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Diabetes Prevention
Keywords: Diabetes Prevention; Lifestyle Intervention; African American Families

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Family-Based intervention (Active Comparator): Families randomized to the Standard Family-based Intervention will receive three-month family YMCA memberships, one orientation training session, access to available equipment and programming at the YMCA, and receive diabetes educational materials from the "Power to Prevent" curriculum via email. Based on our previous experience with AA adults, the investigators anticipate that all families will have access to email either at home or at work. Educational materials will be mailed to families without access to email. The study will also maintain contact with participants by sending holiday and birthday cards, as well as postcard reminders of scheduled data collection visits.
  Interventions: Behavioral: Standard Family-Based intervention
- Lifestyle Intervention (Experimental): The lifestyle intervention for adults will involve a dietary weight loss program and an increase in caloric expenditure through moderate PA. Parents will be encouraged to decrease caloric intake in a sound manner to produce a total weight loss of 5%. The PA component will be to promote an increase in family home-based activity.
  Children. The study will promote healthy eating behaviors, rather than restrictive eating plans with caloric restrictions.
  Interventions: Behavioral: Lifestyle Intervention

INTERVENTIONS:
Behavioral: Lifestyle Intervention — Family-based group lifestyle intervention
  Arms: Lifestyle Intervention
Behavioral: Standard Family-Based intervention — Comparison intervention
  Arms: Standard Family-Based intervention

SUMMARY:
In response to the growing threat of obesity on the health of American children, specifically African American children, the investigators propose to develop a program to educate and motivate African American families to improve health behavior for obesity reduction and diabetes prevention. This project will be unique in its partnership with local YMCAs and its use of Family Health Coaches from the YMCAs who will work one-on-one with participating families. The investigators feel this program will benefit all members of the families who are enrolled and will encourage all members to participate though the study will target one parent and one child who is 8 to 10 years old.

DETAILED DESCRIPTION:
The investigators' long-term research goal is to translate the Diabetes Prevention Program (DPP) in community-based settings for overweight/obese African American (AA) families at risk for Type 2 Diabetes Mellitus (T2DM). Intensive lifestyle approaches addressing physical activity, healthy eating patterns, and stress management are established methods for reducing obesity and risk of T2DM for adults (Knowler, 2002; Tuomilehto et al, 2001; Pan et al, 1997). But, minimal evidence exists that this knowledge has been translated in sustainable settings or in a manner that acknowledges the influences of daily life on motivation and family self-efficacy for changes in nutrition and physical activity. The study proposes to adapt these components for AA families through the use of "family coaches", one-on-one intervention sessions through supervised individualized physical activity, and tailoring intervention strategies for individual families. Utilizing a family systems approach, each component will be delivered using brief motivational strategies that will target self-efficacy and motivational readiness. This four month, two-arm randomized clinical trial, Parents and Children Together Preventing Diabetes (PACT PD) will test the central hypothesis that, relative to a control condition, a "family health coaching" intervention focused on nutrition and physical activity using brief motivational strategies will improve targeted dietary and physical activity behaviors in overweight/obese AA parents and their overweight/obese 8-10 year old children, (N=50 families) all of whom are at risk for T2DM diabetes. This study will test the feasibility and acceptability of training YMCA fitness staff to utilize brief motivational interviewing and serve as "family health coaches". This study will evaluate the early efficacy of the newly translated, family-based diabetes prevention intervention in improving anthropometric measures of BMI (primary outcome) and waist circumference, physical activity and dietary intake, and family functioning (secondary outcomes) and intervention fidelity, feasibility and acceptability of participants. Further, the study will assess the acceptability and feasibility of booster interventions for motivation maintenance and potential for long-term retention and intervention success in the subsequent R18 application. This study will provide critical information regarding the early effectiveness of an innovative, family-based, behavioral intervention for the prevention of T2DM specifically translated for AA families. This study is funded by the National Institutes for Diabetes and Digestive and Kidney Disorders.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass index (One overweight/obese parent (25 kg/m2 <BMI<40 kg/m2 and one overweight/obese child (at or above the 85th% of age-and gender- specific BMI)
* Parental HbA1c levels (pre-diabetes = 5.7 - 6.4%)
* Parent and their child age 8-10

Exclusion Criteria:

* Clinical history of T2DM
* On glucose-lowering drugs
* Currently participating in a supervised weight loss program
* Pregnant or Breastfeeding
* Has conditions limiting participation in the interventions
* Has undergone weight loss surgery
* Unwilling to accept randomization
* Plans to live outside the general area in the next 6 months

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-03; Primary Completion 2015-04-16 (Actual); Study Completion 2015-04-16 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | 12 weeks and 16 weeks.
  The study will assess change in body mass index in both parents and children at 2 post-randomization time points. We will compare these with baseline BMI.

SECONDARY OUTCOMES:
Waist Circumference | 12 weeks and 16 weeks.
Physical activity | 12 weeks and 16 weeks
  The study will measure physical activity in parents and children by accelerometry.
Dietary Intake | 12 weeks and 16 weeks
  The study will use BLOCK measures for both children and parents to assess dietary intake.
Blood Pressure | 12 weeks and 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Beech, DrPH, Principal Investigator — Wake Forest University; Edward Ip, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States